CLINICAL TRIAL: NCT01364363
Title: Allogeneic Hematopoietic Progenitor Cell Transplantation From Unrelated Donors
Brief Title: Unrelated Donor Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIRB#13-6190
Record Dates: First submitted 2011-04-04; First posted 2011-06-02 (Estimated); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Severe Aplastic Anemia; Paroxysmal Nocturnal Hemoglobinuria; Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndromes; Myeloproliferative Syndromes; Chronic Myelogenous Leukemia; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Multiple Myeloma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Large Granulocytic Leukemia
Keywords: Transplant; Allogeneic; Allogeneic transplant; Unrelated donor transplant; MUD; HSCT; Stem cell transplant
MeSH Terms: conditions — Anemia, Aplastic; Hemoglobinuria, Paroxysmal; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hodgkin Disease; Lymphoma, Non-Hodgkin; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Transplantation, Homologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Total Body Irradiation/VP16 (Other): Acute Leukemias, Myelodysplastic syndromes
  Interventions: Procedure: Allogeneic transplantation
- Cytoxan/Total Body Irradiation (Other): Chronic Leukemias, Bone Marrow Failure States, Lymphomas, Hodgkin's Disease
  Interventions: Procedure: Allogeneic transplantation
- Busulfan/Cytoxan (Other): Acute Leukemia, Myelodysplastic syndromes, Chronic Leukemias, Bone Marrow Failure states
  Interventions: Procedure: Allogeneic transplantation
- BEAM (BCNU, etoposide, Ara-C, melphalan) (Other): Lymphomas, Hodgkin's Disease
  Interventions: Procedure: Allogeneic transplantation
- Total Lymphoid Irradiation (Other): For patients with Multiple Myeloma, or prior autologous transplantation, or age in excess of 55
  Interventions: Procedure: Allogeneic transplantation
- Cladribine/Melphalan (Other): For patients with Multiple Myeloma, or prior autologous transplantation, or age in excess of 55
  Interventions: Procedure: Allogeneic transplantation
- FLAG (fludarabine, Ara-C, G-CSF) (Other): For patients undergoing a second allogeneic transplant
  Interventions: Procedure: Allogeneic transplantation

INTERVENTIONS:
Procedure: Allogeneic transplantation — Allogeneic transplantation with matched unrelated donors
  Other Names: MUD transplant

SUMMARY:
The purpose of this study is to provide an opportunity for patients with malignancies or bone marrow failure states who lack a suitable sibling donor to undergo allogeneic hematopoietic progenitor cell transplantation using cells from unrelated individuals or cord blood registries.

DETAILED DESCRIPTION:
same

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of Age
* < 70 years
* ECOG performance status 0, 1 or 2
* Left Ventricular Ejection Fraction > 30%
* Creatinine clearance > 40ml/min
* Transaminases < 2X normal
* Total bilirubin < 2X normal
* HIV seronegativity
* Weight < 70kg for cord blood transplantation
* Ability to cover the cost of the transplant, necessary medications, and transportation/housing.
* Caregiver must be available while outpatient

Exclusion Criteria:

* Greater than one antigen mismatch at HLA-A, B, C or DR plus one allele mismatch at HLA-A, B, C or DR

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Bone Marrow and Peripheral Blood Chimerism | 30 days post-transplant
  Percent of donor and host cells in peripheral blood and bone marrow will be measured by short tandem repeat (STR) testing and/or standard cytogenetic testing.
Bone Marrow and Peripheral Blood Chimerism | 100 days post-transplant
  Percent of donor and host cells in peripheral blood and bone marrow will be measured by short tandem repeat (STR) testing and/or standard cytogenetic testing.
Bone Marrow and Peripheral Blood Chimerism | 365 days post-transplant
  Percent of donor and host cells in peripheral blood and bone marrow will be measured by short tandem repeat (STR) testing and/or standard cytogenetic testing.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W. Andrey, MD, Principal Investigator — Scripps Clinic Medical Group
Locations (1):
- Scripps Green Hospital, La Jolla, California, United States